CLINICAL TRIAL: NCT07055451
Title: A Phase 1b Study to Evaluate the Safety and Pharmacokinetics of Bictegravir/Emtricitabine/Tenofovir Alafenamide (B/F/TAF) in Neonates Exposed to HIV-1
Brief Title: Study of Bictegravir/Emtricitabine/Tenofovir Alafenamide in Newborns Exposed to HIV
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-380-5578
Record Dates: First submitted 2025-06-27; First posted 2025-07-09 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Group A of B/F/TAF (Experimental): Full-term neonate participants, who are exposed to HIV-1 but uninfected, with a weight of ≥ 2.5 kg at birth and their mothers will be assigned to Cohort 1 Group A to evaluate a different pharmacokinetic (PK) sampling scheme than Cohort 1 Group B.
  Neonate participants will receive a single dose of B/F/TAF fixed-dose combination 1.88/7.5/0.94 mg tablet for oral suspension administered along with 1 antiretroviral as standard of care postnatal prophylaxis at both Visits 1 and 3.
  Interventions: Drug: B/F/TAF
- Cohort 1: Group B of B/F/TAF (Experimental): Once enrollment in Cohort 1 Group A is completed, full-term neonate participants, who are exposed to HIV-1 but uninfected, with a weight of ≥ 2.5 kg at birth and their mothers will be assigned to Cohort 1 Group B to evaluate a different PK sampling scheme than Cohort 1 Group A.
  Participants will receive a single dose of B/F/TAF fixed-dose combination 1.88/7.5/0.94 mg tablet for oral suspension administered along with 1 antiretroviral as standard of care postnatal prophylaxis at both Visits 1 and 3.
  Interventions: Drug: B/F/TAF

INTERVENTIONS:
Drug: B/F/TAF — Tablet for oral suspension administered

SUMMARY:
The goal of this clinical study is to learn more about the study drug, Bictegravir/Emtricitabine/Tenofovir Alafenamide (B/F/TAF), safety, tolerability, and pharmacokinetics (how B/F/TAF is absorbed, modified, distributed, and removed from the body of the participants) in neonates exposed to human immunodeficiency virus type 1 (HIV-1).

The primary objective of this study is to evaluate the safety and plasma pharmacokinetics (PK) (how B/F/TAF is absorbed, modified, distributed, and removed from the body of the participants) of B/F/TAF tablet for oral suspension (TOS) in full-term neonates exposed to HIV-1 but uninfected.

ELIGIBILITY:
Key Inclusion Criteria:

Mother inclusion criteria:

* Be on standard of care (SOC) antiretroviral therapy for human immunodeficiency virus type 1 (HIV-1) treatment.
* Have confirmed HIV-1 infection based on positive test results obtained from medical records.

Neonate inclusion criteria:

* Be born at term (≥ 37.0 weeks gestational age).
* Be able to take oral medication.
* Be ≤ 120 hours of life at enrollment.
* Have a birth weight ≥ 2.5 kg.
* Is receiving or plans to receive HIV-1 SOC prophylaxis regimen with 1 antiretroviral (ARV) to prevent perinatal transmission.

Key Exclusion Criteria:

Mother exclusion criteria:

* Has a maternal-fetal blood group incompatibility identified by clinically relevant antibody that can cause hemolytic diseases of the neonate.
* Is breastfeeding or plans to breastfeed while on bictegravir (BIC) or emtricitabine (FTC) containing regimen. Mothers on BIC or FTC containing regimen, but not breastfeeding, can be enrolled in the study.

Neonate exclusion criteria:

* Had prior or expected to require blood exchange transfusion.
* Is receiving or plans to receive any component of B/F/TAF or dolutegravir as part of their SOC ARV prophylaxis regimen.
* Has a documented positive HIV-1 nucleic acid test.
* Has Grade 2 or higher aspartate aminotransferase, total bilirubin, hemoglobin, platelets or creatinine. Has Grade 1 or higher alanine aminotransferase.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Max Age: 120 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAs) Though Week 8 After Neonate Birth | First dose date up to 8 Weeks
Percentage of Participants Experiencing Treatment-emergent Laboratory Abnormalities Through Week 8 After Neonate Birth | First dose date up to 8 Weeks
Pharmacokinetic (PK) parameters for Bictegravir (BIC): AUCinf | Predose up to 72 hours postdose
  AUCinf is defined as area under the concentration versus time curve extrapolated to infinite time.
PK parameters for BIC: AUClast | Predose up to 72 hours postdose
  AUClast is defined as the area under the concentration versus time curve from time zero to the last quantifiable concentration.
PK parameters for BIC: AUC0-24h | Predose up to 24 hours postdose
  AUC0-24h is defined as the partial area under the concentration versus time curve from time 0 to time 24 hours.
PK parameters for BIC: Cmax | Predose up to 72 hours postdose
  Cmax is defined as the maximum observed concentration of drug.
PK parameters for BIC: Tmax | Predose up to 72 hours postdose
  Tmax is defined as the time (observed time point) of Cmax.
PK parameters for BIC: Cmin | Predose up to 72 hours postdose
  Cmin is defined as the minimum observed concentration of drug.
PK parameters for BIC: C24h | At 24 hours postdose
  C24h is defined as the concentration of drug at time 24 hours.
PK parameters for BIC: t1/2 | Predose up to 72 hours postdose
  t1/2 is defined as the terminal elimination half-life.
PK parameters for BIC: Apparent CL/F | Predose up to 72 hours postdose
  Apparent CL/F is defined as the apparent total body clearance for extravascular administration.
PK parameters for BIC: Apparent Vz/F | Predose up to 72 hours postdose
  Apparent Vz/F is defined as the apparent volume of distribution based on the terminal phase.

SECONDARY OUTCOMES:
PK Parameters for Emtricitabine (FTC), and Tenofovir (TFV): AUCinf | Predose up to 72 hours postdose
  AUCinf is defined as the area under the concentration versus time curve extrapolated to infinite time.
PK parameters for FTC, TAF, and TFV: AUClast | Predose up to 72 hours postdose
  AUClast is defined as the area under the concentration versus time curve from time zero to the last quantifiable concentration.
PK parameters for FTC, TAF, and TFV: AUC0-24h | Predose up to 24 hours postdose
  AUC0-24h is defined as the partial area under the concentration versus time curve from time 0 to time 24 hours.
PK parameters for FTC, TAF, and TFV: Cmax | Predose up to 72 hours postdose
  Cmax is defined as the maximum observed concentration of drug.
PK parameters for FTC, TAF, and TFV: Tmax | Predose up to 72 hours postdose
  Tmax is defined as the time (observed time point) of Cmax.
PK parameters for FTC, TAF, and TFV: Cmin | Predose up to 72 hours postdose
  Cmin is defined as the minimum observed concentration of drug.
PK parameters for FTC, TAF, and TFV: C24h | At 24 hours postdose
  C24h is defined as the concentration of drug at time 24 hours.
PK parameters for FTC, TAF, and TFV: t1/2 | Predose up to 72 hours postdose
  t1/2 is defined as the terminal elimination half-life.
PK parameters for FTC and TAF: Apparent CL/F | Predose up to 72 hours postdose
  Apparent CL/F is defined as the apparent total body clearance for extravascular administration.
PK parameters for FTC and TAF: Apparent Vz/F | Predose up to 72 hours postdose
  Apparent Vz/F is defined as the apparent volume of distribution based on the terminal phase.
Mother/Caregiver Reported Acceptability of B/F/TAF tablet for oral suspension (TOS) | First dose date up to 15 days
  Acceptability assessed by a numeric response between numbers 1-5. Higher scores indicate better acceptability.
Mother/Caregiver Reported Palatability of B/F/TAF tablet for oral suspension (TOS) | First dose date up to 15 days
  Palatability assessed by a numeric response between numbers 1-5. Higher scores indicate better palatability.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (7):
- United States (3):
  - Ronald Reagan UCLA Medical Center (inpatient hospital), Los Angeles, California
  - Grady Health System - Ponce de Leon Center, Atlanta, Georgia
  - St Jude Children's Research Hospital, Memphis, Tennessee
- South Africa (4):
  - Family Centre for Research with Ubuntu (FAMCRU), Cape Town
  - Durban International Clinical Research Site, Enhancing Care Foundation, Durban
  - Perinatal HIV Research Unit (PHRU), Gauteng
  - WITS RHI Shandukani Research Centre, Johannesburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT07055451